CLINICAL TRIAL: NCT01738113
Title: Open Versus Closed Kinetic Chain Exercises in Tibial Distraction Osteogenesis by Ilizarov's METHOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Lecturer of Orthopedic Physical therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Youssef1
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Limb Length Discrepancy; Bone Deformity
Keywords: Ilizarov; distraction osteogenesis; Muscle architecture; muscle mechanics; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- open kinetic chain exercise (Experimental): Open kinetic chain exercise
  Interventions: Other: Open Kinetic Chain exercise
- Closed Kinetic chain exercise (Experimental): Closed kinetic chain exercise
  Interventions: Other: Closed kinetic chain exercise

INTERVENTIONS:
Other: Open Kinetic Chain exercise — 1. Hamstrings strengthening exercise
  2. Quadriceps strengthening exercise
  3. Hamstrings stretch
  4. Hip extensors and abductors strengthening
  5. Calf-muscles stretching
  6. Strength exercise of ankle dorsiflexors & plantar flexors
  Arms: open kinetic chain exercise
Other: Closed kinetic chain exercise — 1. Foot sliding from sitting
  2. Seated Toe Raises
  3. Hamstrings and quadriceps co-contraction from sitting
  4. Bridging exercise
  5. Sitting-to-standing
  6. Side-to side, forward and backwards weight shifting
  7. Lunge exercise
  8. Squatting exercise
  9. Standing Toe Raises
  10. Standing Hamstrings Stretch
  Arms: Closed Kinetic chain exercise

SUMMARY:
The Ilizarov external fixator is an external skeletal fixator that is used to stabilize or lengthen the limb bones. Bone lengthen bone occurs through mechanical distraction on the long axis of the bone, thus the method of lengthening is called distraction osteogenesis. This method has been shown successful. Unfortunately, it has also been associated with a substantial number of complications.

Muscle shortening and persistent weakness are among the most common complications seen in this procedure. Muscle shortening usually occurs in strong muscle groups such as the planter flexor muscles, as a result of strength imbalance between the opposing muscle groups. Shortening may persist for more than a year after the removal of the fixator and may require surgical intervention. Fortunately, muscular shortening can be prevented by splinting and physiotherapy in the form of stretching and strengthening exercise and functional training.

The use of different exercises in rehabilitation can help accomplishing different therapeutic goals. Thus, the choice to use one or the other should depend on the desired treatment goals. Weight bearing (CKC) and non weight bearing (OKC) exercise has been incorporated into rehabilitation; however, the effects of these two types of exercises particularly on muscle flexibility and mechanics have never been studied systematically.

Therefore, the purpose of this is to compare the effects of OKC and the CKC exercise on muscle strength, architecture and flexibility.

General Hypothesis:

The use of open kinetic or closed kinetic chain exercises will have no different effects on muscle function or internal organization during tibial distraction osteogenesis by Ilizarov's method Specific hypotheses

1. There will be no difference between the effects of OKC and CKC on muscle flexibility.
2. There will be no difference between the effect of OKC and CKC exercises on muscle strength.
3. There will be no difference between the effect of OKC and CKC on the internal organization of muscle specifically the pennation angle, muscle thickness and fiber length.
4. There will be no difference between the overall of OKC and CKC exercise on the functional performance of patients.

DETAILED DESCRIPTION:
First, personal information and history of each subject will be collected. Then, patients will be informed and receive a full oral explanation of the purpose and procedures of the study before they will be asked to sign an informed consent form.

An initial assessment will be done at the end of latent period (5-7 days) and then every 2 weeks thereafter for a period of 3-5cm distraction or the end of distraction period whatever is earlier.

Patients enrolled in this study will be divided randomly into two groups (A & B). Group A (OKC): will consist of 10 patients receiving open-kinetic- chain exercise program. Group B (CKC) will consist of 10 patients receiving closed-kinetic- chain exercise program.

Initially, each patient will be assessed using the Borg scale to determine the number of strengthening exercise repetitions that patient can carry out. Assessment will be repeated weekly, before the number of repetition is progressed. For stretching exercise, 5 repeat ions will be done each session, in addition patients will be asked to repeat the exercise as a home program exercise. Exercise will be given 3 times weekly, at the University of Benha outpatient clinic, for a period of 3-5 cm of distraction (approximately 8 weeks) or the end of distraction whatever is earlier Exercise for group (A) Knee flexion exercise Patient in supine and gently bend his knee, with keeping the heel in contact with the bed. Bring the heel towards bottom as far as is comfortable .Exercise will be repeated as determined by patient's ability.

Strength the hamstring muscle Patient will be in prone lying position with the knee free out of the bed. Patient will then be asked to bend his knee by making the heel touches his bottom.

Strength quadriceps muscle Patient will sit on the edge of bed or on chair with the thigh supported. Patient will be asked to keep his trunk upright. Then, the knee will be straightened and will be held with the toes pointing to the ceiling for 6 seconds.

Stretch hamstring from sitting:

Patients will assume the long sitting position with their non-operated extremity hanging over the edge of the bed. Patients will then lean forward, grasp his/her forefoot and dorsiflex the ankle while maintaining the knee extended. This position will be maintained for 20-60 seconds before returning to the starting position. The whole exercise will be repeated for 5 times.

Stretch hamstring from prone:

Patients will assume a prone lying position. The legs of the operated limb will be positioned in a neutral rotation and will be allowed to hang freely, over the edge of the bed, by the weight of leg and apparatus as well as by the pulling effect of the gravity. This position will be maintained for duration ranges from 1 minute to as long as tolerated by every individual patient. Patients will also be instructed to assume this position frequently at home during some daily activities e.g. while watching television or reading a book.

Strength hip extensor and abductors:

Patient will be prone with extended knee. Patient will be asked to raise the lower limb upward with the knee extended. For abductor strengthening, the patient will be in a side lying position on the non-operated limb and will be asked to raise the upper limb upwards while the knee is kept straight.

Calf-muscles stretch:

To stretch the gastrocnemius, the patient's heel will be grasped while the knee is extended. Then, the calcaneus will be pulled caudally, with the thumb and fingers of the therapist, before the heads of the metatarsals are gently pushed upwards. The end position will be held for 20-60 seconds before rest is allowed.

Strength exercise for dorsiflexors plantar flexors Patient in long sitting using Theraband one end by his hands and the other end secure around metatarsal bone then the patient will perform plantar flexion against resistance of surgical tubing repeat 10 times.

Exercise for group (B) Wall slides Patient will stand with back against a wall, and feet straight in front of him. Patient then slide down keeping back against the wall, until becoming in a slight sitting position. Slide down only as far as patient feel comfortable. For the first few times patient do this knee exercise, hold the sitting position for a few seconds, then slide back up repeat 10 times.

Foot sliding from sitting While patient is sitting on a smooth surface, the patient pulls the heel of involved leg toward buttocks, flexing the knee as much as tolerable. Hold and straighten leg by sliding heel downward.

Hamstring and quadriceps co-contraction from sitting From a relaxed sitting position with both knees bent to 90 degrees, the patients will be instructed to press firmly on the ground. This exercise will also be done using a stepper machine. Patient was instructed to press rhythmically on the feet plate of a stepper machine, while maintaining the feet in complete contact with the plate, so that heels were vertical.

Bridging exercise:

Patient will assume the crock lying position. In this position, the knees were bent to 30-45 degrees while the feet are completely resting on the supporting surface by placing a firm wedge underneath the feet to accommodate them to the supporting surface. Then, patients will be instructed to raise their lower back and pelvis, while bearing weight on both lower limbs, until the thighs lies in line with pelvis and trunk.

Side-to side, forward and backward weight shifting:

Patient will assume an erect standing position. Both feet will be placed slightly apart with the operated limb placed parallel to, in front of and behind the sound side during side-to-side, forward and backward weight shifting exercise, respectively.

Sitting-to-standing:

Patient will assume a relaxed sitting position. The foot of the affected extremity will be placed initially in front, later, behind the other side. Patient will be instructed to assume the standing positing, while bearing as much weight as they can on their affected extremities.

Lunge exercise:

Patient will assume the forward lunge position. In this position, the affected limb will be placed in front of the other. The distance through which each subject lunged forward will be determined by each individual's leg length as the feet should be about 2 to 3 feet apart, depending on patient's leg length. Then, each subject will move from an upright standing position to the forward lunge position, and back to the starting position.

Squatting exercise:

Patient will be instructed to stand erect, between the parallel bars, with their feet parallel and slightly apart. While maintaining the back erect, they will be instructed to bend both knees slightly then to return back to the erect standing position by pushing against the feet.

Standing Toe Raises:

This exercise is more advanced than the seated toe raise, as it places the entire weight of the body on the exercised leg. Stand upright on both feet Push down through the toes lifting both heels off the ground

Standing Hamstring Stretch:

Patient will stand in front of an elevated surface. Place the operated leg on the surface, Lean forward from the hips until a gentle hamstring stretch is felt on the underside of the thigh. Once a gentle hamstring stretch is felt on the underside of the thigh, hold this position for 30 seconds

ELIGIBILITY:
Inclusion Criteria:

* Referred from an orthopedic surgeon with diagnosis of tibial lengthening or deformity correction by Ilizarov's external fixator.
* unilateral or bilateral tibial distraction osteogenesis.

Exclusion Criteria:

* Patients with Ilizarov due to neurological causes (e.g. poliomyelitis) or other neuromusculoskeletal disease that could affect muscle function and innervations.
* Ankle or knee joints are included in the Ilizarov frame.
* Patients developed neurological complications that interfere with rehabilitation after the application of the Ilizarov apparatus.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
peak isometric strength of the ankle plantar flexors | september 2013 (10 months)
  Then Isometric strength of the ankle plantar flexors will be measured using an isometric test in which the patients push maximally against the plate and the piston of the hand-held dynamometer for four to five seconds. Three measurements will be taken, with only maximum value used for statistical analysis

SECONDARY OUTCOMES:
Ultrasonography for measuring internal muscle structure | September 2013 (10 months)
  For each patient, images of medial gastrocnemius will be taken bilaterally with the ankle joint at neutral position and at maximum plantar flexion, while the subtalar position is neutral. Imaging will be repeated while the muscle is relaxed and contracting by the same radiologist. The recorded scans will be used to measure Pennation angle, muscle thickness and fiber length using computer software
Ankle plantar flexors flexibility | September 2013 (10 months)
  The flexibility of the gastrocnemius and the soleus muscles will be assessed passively with the knee extended and flexed, respectively. Patient will assume the supine lying position during the testing. The investigator will measure the range of ankle dorsiflexion achieved using a digital inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University; Khaled Ayad, PhD, Principal Investigator — Cairo University; Gamal A hosny, PhD, Study Director — Benha University
Locations (1):
- The University of Banha, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aagaard P, Andersen JL, Dyhre-Poulsen P, Leffers AM, Wagner A, Magnusson SP, Halkjaer-Kristensen J, Simonsen EB. A mechanism for increased contractile strength of human pennate muscle in response to strength training: changes in muscle architecture. J Physiol. 2001 Jul 15;534(Pt. 2):613-23. doi: 10.1111/j.1469-7793.2001.t01-1-00613.x. PMID 11454977
- [Background] Aggeloussis N, Giannakou E, Albracht K, Arampatzis A. Reproducibility of fascicle length and pennation angle of gastrocnemius medialis in human gait in vivo. Gait Posture. 2010 Jan;31(1):73-7. doi: 10.1016/j.gaitpost.2009.08.249. Epub 2009 Sep 22. PMID 19775893
- [Background] Aronson J, Harp JH. Mechanical forces as predictors of healing during tibial lengthening by distraction osteogenesis. Clin Orthop Relat Res. 1994 Apr;(301):73-9. PMID 8156700
- [Background] Augustsson J, Esko A, Thomee R, Svantesson U. Weight training of the thigh muscles using closed vs. open kinetic chain exercises: a comparison of performance enhancement. J Orthop Sports Phys Ther. 1998 Jan;27(1):3-8. doi: 10.2519/jospt.1998.27.1.3. PMID 9440034
- [Background] Bohannon RW. Test-retest reliability of hand-held dynamometry during a single session of strength assessment. Phys Ther. 1986 Feb;66(2):206-9. doi: 10.1093/ptj/66.2.206. PMID 3945674
- [Background] Blazevich AJ. Effects of physical training and detraining, immobilisation, growth and aging on human fascicle geometry. Sports Med. 2006;36(12):1003-17. doi: 10.2165/00007256-200636120-00002. PMID 17123325
- [Background] Coglianese DB, Herzenberg JE, Goulet JA. Physical therapy management of patients undergoing limb lengthening by distraction osteogenesis. J Orthop Sports Phys Ther. 1993 Mar;17(3):124-32. doi: 10.2519/jospt.1993.17.3.124. PMID 8472076
- [Background] Caiozzo VJ, Utkan A, Chou R, Khalafi A, Chandra H, Baker M, Rourke B, Adams G, Baldwin K, Green S. Effects of distraction on muscle length: mechanisms involved in sarcomerogenesis. Clin Orthop Relat Res. 2002 Oct;(403 Suppl):S133-45. doi: 10.1097/00003086-200210001-00016. PMID 12394462
- [Background] Dahl MT, Gulli B, Berg T. Complications of limb lengthening. A learning curve. Clin Orthop Relat Res. 1994 Apr;(301):10-8. PMID 8156659
- [Background] Fink B, Krieger M, Strauss JM, Opheys C, Menkhaus S, Fischer J, Ruther W. Osteoneogenesis and its influencing factors during treatment with the Ilizarov method. Clin Orthop Relat Res. 1996 Feb;(323):261-72. doi: 10.1097/00003086-199602000-00036. PMID 8625590
- [Background] Fitch RD, Thompson JG, Rizk WS, Seaber AV, Garrett WE Jr. The effects of the Ilizarov distraction technique on bone and muscle in a canine model: a preliminary report. Iowa Orthop J. 1996;16:10-9. PMID 9129270
- [Background] Ghoneem HF, Wright JG, Cole WG, Rang M. The Ilizarov method for correction of complex deformities. Psychological and functional outcomes. J Bone Joint Surg Am. 1996 Oct;78(10):1480-5. doi: 10.2106/00004623-199610000-00004. PMID 8876574
- [Background] Physiotherapy during Ilizarov fixation. Techniques Orthop; 5(4):61-65, 1990.
- [Background] Green SA. Patient management during limb lengthening. Instr Course Lect. 1997;46:547-54. No abstract available. PMID 9143998
- [Background] Legerlotz K, Smith HK, Hing WA. Variation and reliability of ultrasonographic quantification of the architecture of the medial gastrocnemius muscle in young children. Clin Physiol Funct Imaging. 2010 May;30(3):198-205. doi: 10.1111/j.1475-097X.2010.00925.x. Epub 2010 Feb 23. PMID 20184623
- [Background] Maganaris CN, Baltzopoulos V, Sargeant AJ. In vivo measurements of the triceps surae complex architecture in man: implications for muscle function. J Physiol. 1998 Oct 15;512 ( Pt 2)(Pt 2):603-14. doi: 10.1111/j.1469-7793.1998.603be.x. PMID 9763648
- [Background] Paley D. Problems, obstacles, and complications of limb lengthening by the Ilizarov technique. Clin Orthop Relat Res. 1990 Jan;(250):81-104. PMID 2403498
- [Background] Schep NW, van Lieshout EM, Patka P, Vogels LM. Long-term functional and quality of live assessment following post-traumatic distraction osteogenesis of the lower limb. Strategies Trauma Limb Reconstr. 2009 Dec;4(3):107-12. doi: 10.1007/s11751-009-0070-3. Epub 2009 Nov 24. PMID 19937148
- [Background] Shyam AK, Song HR, An H, Isaac D, Shetty GM, Lee SH. The effect of distraction-resisting forces on the tibia during distraction osteogenesis. J Bone Joint Surg Am. 2009 Jul;91(7):1671-82. doi: 10.2106/JBJS.G.01238. PMID 19571090
- [Background] Ilizarov tension stress
- [Background] The principles of the Ilizarov method
- [Background] Ilizarov GA. The tension-stress effect on the genesis and growth of tissues: Part II. The influence of the rate and frequency of distraction. Clin Orthop Relat Res. 1989 Feb;(239):263-85. PMID 2912628
- [Background] Ilizarov GA. The tension-stress effect on the genesis and growth of tissues. Part I. The influence of stability of fixation and soft-tissue preservation. Clin Orthop Relat Res. 1989 Jan;(238):249-81. PMID 2910611
- [Background] Ilizarov GA. Clinical application of the tension-stress effect for limb lengthening. Clin Orthop Relat Res. 1990 Jan;(250):8-26. PMID 2403497
- [Background] Ilizarov GA, Shchurov VA. [Effect of stretching tension on the biomechanical properties of the muscles, their blood supply and the growth of the leg]. Fiziol Cheloveka. 1988 Jan-Feb;14(1):26-32. No abstract available. Russian. PMID 3169414
- [Background] Ilizarov GA. Some possibilities with our method for treating damage to and disorders of locomotor apparatus. J Craniofac Surg. 1995 Sep;6(5):352-4; discussion 355. doi: 10.1097/00001665-199509000-00002. No abstract available. PMID 9020712